CLINICAL TRIAL: NCT01751763
Title: Investigations of Sorafenib for HCC Patients Who Have Residue Disease After Resection With Curative Intent
Brief Title: Sorafenib for Residue Disease After Resection With Curative Intent
Acronym: SECURE
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16621; NX1218CN (Other: company internal)
Record Dates: First submitted 2012-12-14; First posted 2012-12-18 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — treatment (including dose, duration, modification) decided by the investigator.

SUMMARY:
Radical hepatic resection represents one of the treatment options offering a prospect for cure with 5-year survival rates up to 50%. However, unintentionally, quite a proportion of these "radical resection" actually turned out to be non-radical in nature. For these patients who actually received non-radical resection, their by year survival rates were much lower than those who received radical hepatectomy. In this prospective, non-interventional, multi-center study, we are planning to observe the patient characteristics of Hepatocellular carcinoma (HCC) patients who have residual disease after resection with curative intent, as well as treatment pattern, safety and effectiveness of sorafenib for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed HCC and have residual disease after resection with curative intent and for whom a decision to treat with Sorafenib has been made.

The definitions of non-radical resection are as follows:

Liver tumor rupture or adjacent organ invasion, confirmed by intra-operative or post-operative pathology; Positive resection margin, confirmed by post- operative pathology; Lymph node metastasis confirmed by intra-operative or post- operative pathology; Residue lesion confirmed by post-operative digital subtraction angiography (DSA); Macroscopic/microscopic tumor thrombi of vein and/or bile duct, confirmed intraoperative / post-operative pathology; Number of tumors >=3, confirmed by preoperative radiographic inspection (CT, MRI or BUS), intraoperative BUS, or post-operative pathology.

AFP alpha fetoprotein(AFP) remains higher than Upper Limits of Normal (according to local lab's range), confirmed by local laboratory test at least 2 months after surgery.

* Confirmation of complete response (no visible residual tumor), on the eligibility scan (CT or MRI) by local radiological review, performed >2 weeks after surgery;
* Patients must be followed up regularly after surgery (time interval and method based on physician's daily practice), have no documented tumor recurrence by eligibility scan (CT or MRI) before Sorafenib treatment;
* Patients must have physically/mentally recovered from surgery and considered to be able to tolerant Sorafenib therapy, by investigator's judgment;

Exclusion Criteria:

* The approved local product label must be followed for the exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCC patients with residue disease after resection with curative intent
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2013-07-09 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-09-08 (Actual)

PRIMARY OUTCOMES:
Patient characteristics: demographic, baseline characteristic, HCC diagnosis, prior HCC treatment, tumor status at operation, hepatic resection, time interval between surgery and Sorafenib, postoperative anti HCC treatment if any, past medical history | up to 1 year
Treatment pattern of Sorafenib: duration and doses of Sorafenib, dose modification/discontinuation of Sorafenib, concomitant anti-cancer therapy, treatment after observed radiological recurrence. | up to 3 years

SECONDARY OUTCOMES:
Number of participants with adverse events( AE) and Serious adverse events(SAE) as a measure of safety and tolerability | up to 3 years
Disease-free survival (DFS) | up to 3 years
Recurrence rate by year | up to 3 years
survival rate by year | up to 3 years
Overall survival (OS) | up to 3 years
Time to recurrence (TTR) | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, China